CLINICAL TRIAL: NCT02727374
Title: Fear to Fall Reduction in Geriatric Patients Who Suffered Previous Falls
Acronym: FFALL_GER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Celedonia Igual, Dr., University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI_UValencia1
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Geriatric Disorder
Keywords: Fear to Fall; Geriatric; Rehabilitation; Psychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXPERIMENTAL (Experimental): Physiotherapy intervention, plus cognitive-behavioural intervention
  Interventions: Other: Physiotherapy intervention; Behavioral: Cognitive-behavioural Intervention
- CONTROL (Active Comparator): Physiotherapy intervention
  Interventions: Other: Physiotherapy intervention

INTERVENTIONS:
Other: Physiotherapy intervention — Physiotherapy intervention consists of conventional exercise program administered to this kind of patients at Hospital Clinico, including strengthening and balance exercises
Behavioral: Cognitive-behavioural Intervention — Psychological treatment consists of group talks to treat the fear to fall
  Arms: EXPERIMENTAL

SUMMARY:
Fear to fall has been proven to be a risk factor affecting those geriatric patients who have previously suffered a fall. In this work it is assessed the effectiveness of a physiotherapy and psychological combined intervention, aimed at reducing the fear to fall in the aforementioned patients

DETAILED DESCRIPTION:
One of the main consequences of falling is the fear to fall again. This involves changes in the elderly behaviour which leads to a reduction of the physical activity, higher need of cares, reduction of the quality of life and risk of social isolation. In this framework, this works is aimed at performing a treatment to reduce the fear to fall in those geriatrics patients with previous falls, based on the combination of physical activity, health education and cognitive-behavioural psychological treatment targeted to this effect. The reason is that literature points at combined treatment use to present higher effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older people
* Looking for Physiotherapy attendance
* Patients who have suffered at least one fall episode
* Patients with fear of falling

Exclusion Criteria:

* Some cognitive affection that may affect the intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Fear Related Psychological Concerns (Falls) | Prospective change from baseline to end of intervention (8 weeks)
  Assessed in terms of the Falls Efficacy Scale International (FES-I) results
Fear Related Psychological Concerns (Balance) | Prospective change from baseline to end of intervention (8 weeks)
  Assessed in terms of the Activities-Specific Balance Confidence (ABC) scale results
Fear Related Psychological Concerns (Fear) | Prospective change from baseline to end of intervention (8 weeks)
  Assessed in terms of the Visual Analog Scale results (0-10)

SECONDARY OUTCOMES:
Risk of Falling | Prospective change from baseline to end of intervention (8 weeks)
  Assessed in terms of the Timed up & Go test
Center Epidemiological Studies Depression Scale | Prospective change from baseline to end of intervention (8 weeks)
  This is a measurement scale of depression
Ryff Scale | Prospective change from baseline to end of intervention (8 weeks)
  It is a scale for measuring psychological well-being

CONTACTS AND LOCATIONS:
Overall Officials: Celedonia Igual, Professor, Principal Investigator — University of Valencia; Jose M Blasco, PhD, Study Director — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes